CLINICAL TRIAL: NCT01971502
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of BI 1060469 in Healthy Male Volunteers (Single-blind, Placebo-controlled, Randomised, Partly Fixed-sequence, Parallel Group Design) and Effect of Food on the Bioavailability of BI 1060469 (Open-label, Randomised, Two-way Cross-over)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses and Effect of Food on the Bioavailability of BI 1060469
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1333.1; 2013-001475-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-08; First posted 2013-10-29 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 1060469 single rising dose part (Experimental): single rising doses given as tablet
  Interventions: Drug: Placebo to BI 1060469; Drug: BI 1060469
- BI 1060469 food effect part (Experimental): given as tablet fasted and fed
  Interventions: Drug: BI 1060469

INTERVENTIONS:
Drug: Placebo to BI 1060469 — single rising doses
  Arms: BI 1060469 single rising dose part
Drug: BI 1060469 — food effect
  Arms: BI 1060469 food effect part
Drug: BI 1060469 — single rising doses
  Arms: BI 1060469 single rising dose part

SUMMARY:
The objective of the single rising dose part (SRD) is to investigate safety, tolerability, pharmacokinetics, and pharmacodynamics of single rising doses of BI 1060469 in healthy male subjects. The objective of the food effect part (FE) is to investigate the relative bioavailability of BI 1060469 tablets in healthy male subjects in fed or fasted state.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, and clinical laboratory tests
2. Age within the range of 18 to 50 years
3. Body mass index within the range of 18.5 and 29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and judged clinically relevant by the investigator. Pulse rate outside the range of 50-90 bpm or blood pressure outside the ranges of 90-140 for systolic and 50-90 mmHg for diastolic blood pressure if confirmed by repeat measurement.
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. In the SRD: serum creatinine laboratory value outside the normal range
4. Glomerular filtration rate (GFR) according to CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration)-Formula < 60 ml/ min
5. Current or history of relevant kidney, urinary tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
7. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with drug- related adverse events. | up to 2 weeks

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of BI 1060469 in plasma) | up to 2 weeks
AUC0-infinity (area under the concentration-time curve of BI 1060469 in plasma over the time interval from 0 extrapolated to infinity) | up to 2 weeks
AUC0-tz (area under the concentration-time curve of BI 1060469 in plasma over the time interval from 0 up to the last quantifiable data point) | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1333.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany